CLINICAL TRIAL: NCT01539525
Title: Screening to Augment Referral to Treatment- Project START
Acronym: ProjectSTART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kimberly Yonkers, Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1005006785; R01DA027194 (NIH)
Record Dates: First submitted 2011-08-03; First posted 2012-02-27 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Alcohol Abuse; Tobacco Use Disorder; Marijuana Abuse; Substance-Related Disorders
MeSH Terms: conditions — Alcoholism; Tobacco Use Disorder; Marijuana Abuse; Substance-Related Disorders | interventions — Motivational Interviewing; Therapeutics

STUDY DESIGN:
Masking Description: Participants received a behavioral intervention that could not be masked. Outcome data were self report and urine tests rom the participants.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Motivational Interview (Experimental): Motivational interview provided by a clinical research nurse or physician.
  Interventions: Behavioral: Motivational Interview
- Motivational Interview-Electronic (Active Comparator): Motivational Interview provided by an interactive computer program.
  Interventions: Behavioral: Motivational Interview
- Treatment as Usual (Placebo Comparator): No intervention- resource list provided.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Motivational Interview — Motivational Interview provided by either a Nurse or Computer
  Arms: Motivational Interview; Motivational Interview-Electronic
Other: Treatment as Usual — Subjects given a brochure listing relevant recovery resources in the local area.
  Arms: Treatment as Usual

SUMMARY:
The investigators propose to use obstetric-gynecological clinics to conduct a randomized clinical trial that would compare two SBIRTS (Screening, Brief Intervention, Referral and Treatment), delivered either by a trained nurse or by computer, to usual care (a control condition). As part of this trial, the investigators will include outcomes that allow us to assess the cost effectiveness of these three conditions.

DETAILED DESCRIPTION:
Aim 1: To assess whether SBIRT, based upon motivational interviewing and delivered either by computer or a trained nurse, leads to decreased use of a subject's primary drug of abuse.

Hypothesis #1a: Referrals based upon motivational principles and delivered by computer, as compared to usual care (health brochure with treatment resources), will lead to greater reductions in a woman's primary substance of abuse.

Hypothesis #1b: Referrals based upon motivational principles and delivered by nurse, as compared to usual care (health brochure with treatment resources), will lead to greater reductions in a woman's primary substance of abuse.

Aim 2: To determine whether SBIRT based upon motivational interviewing and delivered either by computer or by a nurse will promote substance abuse treatment utilization for the primary drug of abuse.

Hypothesis #2a: Treatment utilization (eg. treatment initiation, attendance, use of quit-line or medication) will be higher if a woman receives the computer delivered brief intervention than if she receives usual care only.

Hypothesis #2b: Treatment utilization (eg. treatment initiation, attendance, use of quit-line or medication) will be higher if a woman receives the nurse delivered brief intervention than if she receives usual care only.

Secondary Aim 3: To evaluate whether SBI leads to a decrease in HIV/AIDS risk

Hypothesis #3: Rates of sexually transmitted diseases, injection drug use and risky sexual behavior will be lower at follow up for subjects who receive either computer or a nurse delivered brief intervention than usual care subjects.

Secondary Aim 4: To compare the relative cost-effectiveness of the three interventions.

Hypothesis #4a: Screening and usual care will be the most cost-effective intervention method when the value of an additional unit of effect for the given individual's outcome is relatively low.

Hypotheses #4b: Screening, and a brief intervention delivered by computer, will be the most cost-effective treatment method when the value of an additional unit of effect is relatively high.

Hypotheses #4c: Screening, and a brief intervention delivered by a nurse, will be less cost-effective than a brief intervention delivered by computer.

ELIGIBILITY:
Inclusion Criteria:

In order to participate, women must meet the following criteria:

1. Are non-pregnant and meet ASSIST criteria for at least moderate risk for alcohol (≥11) or drug (≥4) abuse or dependence (tobacco or illicit drugs, including cocaine, opiates, methamphetamine, marijuana or a prescription drug used in a medically inappropriate manner).
2. Are pregnant and meet ASSIST criteria for at least mild to moderate risk for alcohol (≥6) or drug (≥4) abuse or dependence (alcohol, tobacco, an illicit drug, or a prescription drug in a medically inappropriate manner). We define pregnant women who use alcohol or drugs at least monthly in the last 90 days as eligible because alcohol and many of the other substances (eg. tobacco) are teratogens and use in pregnancy would be consistent with a diagnosis of abuse ("recurrent use in situations in which it is physically hazardous"). This level of use in pregnancy also indicates a greater likelihood of problematic substance use.
3. Have used their primary substance at least once within the prior 28 days.
4. Are aged 18 or more. We include participants who are aged 18 or older because parents may not be available at screening to provide consent for non-pregnant participants and subjects may not wish to disclose drug or alcohol abuse to a parent.

Exclusion Criteria:

Women are ineligible if they have any of the following criteria:

1. Are unable to speak English.
2. Are incarcerated or at risk of incarceration. The YNHH Women's Center provides care to incarcerated women. These individuals as well as those at risk of incarceration are excluded because incarceration precludes their ability to seek specialty drug or alcohol abuse treatment (a dependent measure).
3. Have a cognitive disorder that would impair their ability to provide informed consent or provide accurate information.
4. Require immediate hospitalization because of general medical needs or due to active suicidal or homicidal ideation or other behavioral health problems. We exclude individuals who are in need of immediate hospitalization because hospitalization will render it more difficult for them to immediately follow-up on a referral and because providers, rather than subjects, may be making the decision to initiate treatment. Hospitalization would also potentially force women who smoke to initiate treatment for tobacco addiction.
5. Are currently participating or have participated in drug abuse treatment, including self-help interventions (eg. 12 step facilitation, smoking cessation interventions), within the last 3 months prior to screening.
6. Are planning to relocate out of the area in the following 6 months. Women who relocate out of the area would be difficult to see for follow up assessments and it would be difficult to confirm treatment attendance in local treatment centers.
7. Have previously participated in this protocol or
8. Are unwilling to participate or accept randomization.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 439 (Actual)
Dates: Start 2011-09-05 (Actual); Primary Completion 2015-01-28 (Actual); Study Completion 2015-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Yonkers, MD, Principal Investigator — Yale University; Steve Martino, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale-New Haven Hospital- York St Campus, New Haven, Connecticut
  - Yale-New Haven Hospital-Chapel St Campus, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No
We will require data request with delineation of variables of interest. Only de-identified data will be released after evaluation of the request

REFERENCES:
- [Derived] Forray A, Martino S, Gilstad-Hayden K, Kershaw T, Ondersma S, Olmstead T, Yonkers KA. Assessment of an electronic and clinician-delivered brief intervention on cigarette, alcohol and illicit drug use among women in a reproductive healthcare clinic. Addict Behav. 2019 Sep;96:156-163. doi: 10.1016/j.addbeh.2019.05.007. Epub 2019 May 8. PMID 31100713
- [Derived] Loree AM, Yonkers KA, Ondersma SJ, Gilstad-Hayden K, Martino S. Comparing satisfaction, alliance and intervention components in electronically delivered and in-person brief interventions for substance use among childbearing-aged women. J Subst Abuse Treat. 2019 Apr;99:1-7. doi: 10.1016/j.jsat.2019.01.007. Epub 2019 Jan 9. PMID 30797381

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were women (non-pregnant and pregnant) presenting for outpatient reproductive healthcare in an urban academic hospital-based clinic. Data collection occurred between April 20, 2011 and January 28, 2015.
Groups:
- Motivational Interview-Nurse: Motivational interview provided by a clinical research nurse or physician.
  Motivational Interview: Motivational Interview provided by either a Nurse or Computer
- Motivational Interview-Computer: Motivational Interview provided by an interactive computer program.
  Motivational Interview: Motivational Interview provided by either a Nurse or Computer
- Treatment as Usual: No intervention- resource list provided.
  Resource brochure: Subjects given a brochure listing relevant recovery resources in the local area.
Period: Overall Study
Arm/Group | Motivational Interview-Nurse | Motivational Interview-Computer | Treatment as Usual
Started | 145 | 143 | 151
Completed | 125 | 127 | 134
Not Completed | 20 | 16 | 17
Not completed — Lost to Follow-up | 19 | 12 | 11
Not completed — Withdrawal by Subject | 0 | 3 | 2
Not completed — Protocol Violation | 1 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Interview | Motivational Interview-Electronic | Treatment as Usual | Total
Number analyzed (Participants) | 145 | 143 | 151 | 439
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (109) | 34.6 (10.3) | 34.4 (12.0) | 34.2 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 143 | 151 | 439
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Afican-American, non-Hispanic | 102 | 93 | 98 | 293
  Caucasian-American, non-Hispanic | 19 | 16 | 23 | 58
  Hispanic | 19 | 22 | 24 | 65
  Other race/ethnicity | 5 | 12 | 6 | 23
Marital Status [Number; unit: participants]
  Married/living with partner | 70 | 54 | 73 | 197
  Other living situation | 75 | 89 | 78 | 242
Pregnant [Number; unit: participants]
  Pregnant | 27 | 24 | 29 | 80
  Not pregnant | 118 | 119 | 122 | 359
Education [Number; unit: participants]
  Some high school or less | 46 | 48 | 52 | 146
  High school graduate | 64 | 60 | 57 | 181
  Beyond high school | 35 | 33 | 42 | 110
  missing | 0 | 2 | 0 | 2
Employment status [Number; unit: participants]
  Full-time | 18 | 28 | 20 | 66
  Part-time | 24 | 26 | 32 | 82
  Not working | 103 | 89 | 99 | 291
Primary Substance [Number; unit: participants]
  Nicotine | 81 | 80 | 90 | 251
  Alcohol | 15 | 23 | 13 | 51
  Cannabis | 32 | 27 | 31 | 90
  Other illicit drug | 17 | 13 | 17 | 47
Primary substance use [Mean (Standard Deviation); unit: days per month] | 23.2 (8.3) | 23.7 (7.7) | 24.2 (7.7) | 23.7 (7.9)
Any substance use [Mean (Standard Deviation); unit: days per month] | 26.0 (5.5) | 25.4 (6.2) | 25.7 (6.1) | 25.7 (5.9)
Substance Use Disorders [Number; unit: participants]
  Nicotine | 81 | 80 | 90 | 251
  Alcohol | 15 | 23 | 13 | 51
  Cannabis | 32 | 27 | 31 | 90
  Other illicit drug | 17 | 13 | 17 | 47
Alcohol, Smoking, and Substance Involvement Screening Test Score [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0 to 39, with higher scores indicating greater need for more intensive intervention. Scores are for primary substance.
  units on a scale | 22.5 (8.1) | 22.8 (8.5) | 22.2 (8.1) | 22.5 (7.9)
Fagerstrom Test for Nicotine Dependence Score [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0 to 10, with higher scores indicating higher levels of nicotine dependence.
  units on a scale | 3.8 (2.7) | 3.6 (2.8) | 3.9 (2.7) | 3.9 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Days Per Month of Primary Substance Use
Description: Participants completed a timeline followback at each assessment, reporting days of primary substance use. Outcomes reported are raw means and standard deviations.
Time Frame: 7 non-overlapping monthly intervals from baseline to month 6
Measure: Mean (Standard Deviation); unit: days per month
Arm/Group | Motivational Interview-Nurse | Motivational Interview-Computer | Treatment as Usual
Number analyzed (Participants) | 145 | 143 | 151
days per month
  baseline | 23.2 (8.3) | 23.7 (7.7) | 24.2 (7.7)
  Month 1 | 19.3 (11.2) | 19.7 (11.2) | 22.8 (8.9)
  Month 2 | 18.7 (11.8) | 17.9 (12.1) | 22.2 (10.1)
  Month 3 | 18.0 (12.0) | 17.8 (11.9) | 21.4 (10.6)
  Month 4 | 18.0 (12.2) | 16.8 (12.3) | 20.0 (11.4)
  Month 5 | 17.6 (12.5) | 16.3 (12.6) | 19.7 (11.4)
  Month 6 | 17.0 (12.3) | 16.2 (12.5) | 19.1 (11.8)
Statistical Analysis 1: Comparison: Motivational Interview-Nurse vs Motivational Interview-Computer vs Treatment as Usual; Differences in days/month of primary substance use over time between treatment groups were examined using generalized estimating equations (GEE). We specified a negative binomial distribution to account for overdispersion in days/month of primary substance use, a log link function, and a first-order autoregressive working correlation structure. β coefficients were estimated using quasi-likelihood estimation methods and sandwich/empirical standard errors were calculated; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equation; adjusted for stratifying variables- primary substance and pregnancy status; Slope = -0.078, 95% CI 2-sided [-0.118 to -0.038], Standard Error of Mean 0.020 — Parameter estimated is the linear effect of time (in months)
Statistical Analysis 2: Comparison: Motivational Interview-Nurse vs Motivational Interview-Computer vs Treatment as Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.066, Generalized Estimating Equation; adjusted for stratifying variables- primary substance and pregnancy status; Slope = 0.005, 95% CI 2-sided [-0.0004 to 0.011], Standard Error of Mean 0.003 — Parameter estimated is the quadratic effect of time (in months)
Statistical Analysis 3: Comparison: Motivational Interview-Nurse vs Motivational Interview-Computer vs Treatment as Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.038, Generalized Estimating Equation — P-value adjusted for multiple comparisons using Holm's step-down multiple testing procedure. The a priori threshold for statistical significance was p < 0.05; adjusted for stratifying variables- primary substance and pregnancy status; Slope = -0.078, 95% CI 2-sided [-0.151 to -0.004], Standard Error of Mean 0.034 — Estimated parameter is treatment x linear time interaction term coefficient- Motivational Interview- Nurse vs. Treatment as Usual
Statistical Analysis 4: Comparison: Motivational Interview-Nurse vs Motivational Interview-Computer vs Treatment as Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.008, Generalized Estimating Equation — P-value adjusted for multiple comparisons using Holm's step-down multiple testing procedure. The a priori threshold for statistical significance was p < 0.025; adjusted for stratifying variables- primary substance and pregnancy status; Slope = -0.090, 95% CI 2-sided [-0.157 to -0.023], Standard Error of Mean 0.034 — Estimated parameter is treatment x linear time interaction term coefficient- Motivational Interview- Computer vs. Treatment as Usual
Statistical Analysis 5: Comparison: Motivational Interview-Nurse vs Motivational Interview-Computer vs Treatment as Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.031, Generalized Estimating Equation — [p-value comment as in outcome 1, analysis 3]; adjusted for stratifying variables- primary substance and pregnancy status; Slope = 0.011, 95% CI 2-sided [0.001 to 0.022], Standard Error of Mean 0.005 — Estimated parameter is treatment x quadratic time interaction term coefficient- Motivational Interview- Nurse vs. Treatment as Usual
Statistical Analysis 6: Comparison: Motivational Interview-Nurse vs Motivational Interview-Computer vs Treatment as Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.010, Generalized Estimating Equation — [p-value comment as in outcome 1, analysis 4]; adjusted for stratifying variables- primary substance and pregnancy status; Slope = 0.012, 95% CI 2-sided [0.002 to 0.021], Standard Error of Mean .0005 — Estimated parameter is treatment x quadratic time interaction term coefficient- Motivational Interview- Computer vs. Treatment as Usual

2. Primary Outcome: Treatment Utilization
Description: Treatment utilization assessed via participant self-report at each follow-up interview, and with the exception of self-help groups, verified with providers. We also reviewed the medical record for use of medication indicative of treatment (e.g., nicotine replacement therapy).
Time Frame: baseline to 6 months
Measure: Number; unit: participants
Arm/Group | Motivational Interview-Nurse | Motivational Interview-Computer | Treatment as Usual
Number analyzed (Participants) | 145 | 143 | 151
participants
  utilized treatment | 39 | 39 | 43
  no tretment | 106 | 104 | 108
Statistical Analysis 1: Comparison: Motivational Interview-Nurse vs Motivational Interview-Computer vs Treatment as Usual; Test type: Superiority or Other; p = 0.810, Regression, Logistic; adjusted for stratifying variables- primary substance and pregnancy status; Odds Ratio (OR) = 0.931, 95% CI 2-sided [0.559 to 1.551] — Estimated odds ratio is for Motivational Interview- Nurse vs. Treatment as Usual
Statistical Analysis 2: Comparison: Motivational Interview-Nurse vs Motivational Interview-Computer vs Treatment as Usual; Test type: Superiority or Other; p = 0.990, Regression, Logistic; adjusted for stratifying variables- primary substance and pregnancy status; Odds Ratio (OR) = 0.968, 95% CI 2-sided [0.579 to 1.617] — Estimated odds ratio is for Motivational Interview- Computer vs. Treatment as Usual

3. Secondary Outcome: Rates of STDs
Description: rates of incident std's per patient's medical records
Time Frame: baseline to 6 months
Measure: Number; unit: participants
Arm/Group | Motivational Interview-Nurse | Motivational Interview-Computer | Treatment as Usual
Number analyzed (Participants) | 145 | 143 | 151
participants
  Incident case | 8 | 4 | 6
  Non-incident case | 135 | 138 | 152
  Missing | 2 | 1 | 3
Statistical Analysis 1: Comparison: Motivational Interview-Nurse vs Motivational Interview-Computer vs Treatment as Usual; Test type: Superiority or Other; p = 0.465, Regression, Logistic; adjusted for stratifying variables- primary drug and pregnancy status; Odds Ratio (OR) = 1.258, 95% CI 2-sided [0.409 to 3.871] — odds ratio estimate is for Motivational Interview- Nurse vs. Treatment as Usual
Statistical Analysis 2: Comparison: Motivational Interview-Nurse vs Motivational Interview-Computer vs Treatment as Usual; Test type: Superiority or Other; p = 0.490, Regression, Logistic; Odds Ratio (OR) = 0.749, 95% CI 2-sided [0.205 to 2.732] — Odds ratio estimate is for Motivational Interview- Computer vs. Treatment as Usual

4. Secondary Outcome: Mean Cost for Each Intervention
Description: The data table includes the mean cost for implementation of each intervention from the societal perspective. The costs do not include the research costs
Time Frame: 6 months
Population: This outcome was restricted to participants who had a time stamp for their intervention (n=11 were missing) and had all 6 months of follow-up data.
Measure: Mean (Standard Deviation); unit: dollars
Units Other Than Participants: participants
Arm/Group | Motivational Interview | Motivational Interview-Electronic | Treatment as Usual
Number analyzed (Participants) | 145 | 143 | 151
Number analyzed (participants) | 115 | 123 | 133
dollars | 57.56 (16.12) | 21.07 (4.43) | 21.21 (7.3)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Motivational Interview | Motivational Interview-Electronic | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 0/145 | 0/143 | 0/151
Other Adverse Events (participants affected / at risk) | 0/145 | 0/143 | 0/151

LIMITATIONS AND CAVEATS:
Results may not be generalizable to populations differing from population from which sample was drawn.

Outcomes relied upon self-report, although we did try to verify through lab results for substance use and medical records/ provider for treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No